CLINICAL TRIAL: NCT00911625
Title: Glargine Dosing in Hospitalized Patients With Type 2 Diabetes and Renal Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Mary Ann Emanuele, Professor of Medicine, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201463
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes; Renal Insufficiency
Keywords: glargine; glulisine; type 2 diabetes; renal insufficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — Insulin Glargine; insulin glulisine

STUDY DESIGN:
Intervention Model Description: Eligible participants are randomized to one of the two dosing groups using a 1:1 allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.5 units/kg (Active Comparator): Participants randomized to this arm will receive a standard-dose of 0.5 units/kg daily insulin. Half of this dose will be given as glargine and the other half will be given as glulisine.
  Interventions: Drug: 0.5 units/kg daily insulin
- 0.25 units/kg (Experimental): Participants randomized to this arm will receive an experimental dose of 0.25 units/kg daily insulin. Half of this dose will be given as glargine and the other half will be given as glulisine.
  Interventions: Drug: 0.25 units/kg daily insulin

INTERVENTIONS:
Drug: 0.5 units/kg daily insulin — Participants randomized to receive this intervention will receive a standard-dose of 0.5 units/kg daily insulin. Half of this dose will be given as glargine and the other half will be given as glulisine.
  Other Names: Lantus; Apidra
  Arms: 0.5 units/kg
Drug: 0.25 units/kg daily insulin — Participants randomized to receive this intervention will receive an experimental dose of 0.25 units/kg daily insulin. Half of this dose will be given as glargine and the other half will be given as glulisine.
  Other Names: Lantus; Apidra
  Arms: 0.25 units/kg

SUMMARY:
It is imperative to devise easy to follow, yet appropriate, guidelines for insulin use in renal-impaired patients. This will be done by comparing two regimens: 1) glargine once daily plus mealtime glulisine based on weight alone and 2) a predetermined dosing reduction algorithm with glargine/glulisine based on weight with reduction for decreased estimated GFR by MDRD as follows: < 30 ml/min/1.73m2 or on dialysis reduce dose by 50% from weight based calculation.

DETAILED DESCRIPTION:
This study will enroll 180 hospitalized patients with Type 2 diabetes and moderate to end stage renal insufficiency (estimated glomerular filtration rate is < 30 ml/min/1.73m2 or dialysis) in the Chicagoland area. Participants will be randomized into 1 of 2 protocols after hospital admission. Blood glucose levels will be obtained before meals, at bedtime and whenever necessary for any signs or symptoms of hypoglycemia. The primary endpoint will be the percentage of blood glucose levels reaching goal of 80-180mg/dl. A secondary endpoint will be the percentage of hypoglycemic events, defined as blood glucose values < 60 mg/dl. In addition the percentage of glucose levels within the goal range of 80-180mg.dl will be further separated into excellent control (80-140mg/dl) and acceptable control (141-180mg/dl).

The 2 study groups will be:

1. Glargine & glulisine. The total daily insulin dose will be 0.6 units/kg. Half of this will be given as glargine once daily. The other half will be given as glulisine, divided equally between breakfast, lunch, and dinner with correction factor dosing as needed for elevated premeal hyperglycemia.
2. Glargine & glulisine The calculation for the total daily insulin dose will be 0.3 units/kg. Half of this will be given as glargine in the morning. The other half will be given as glulisine, divided equally between breakfast, lunch, and dinner, with correction factor dosing as needed for elevated premeal hyperglycemia.

All oral agents will be discontinued on admission.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus of mor than 1year
* GFR less than 30 ml/min/1.73m2 or dialysis
* Age greater than 18years
* Entry blood glucose (fasting or random) greater than 180mg%

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* New onset hyperglycemia
* Pregnant
* Solid organ transplant within 1 year
* Steroids prednisone greater than 7.5mg/day or equivalent
* Hospital LOS predicted less than 2 days
* Severe liver disease
* Known hypopituitarism or adrenal insufficiency
* Patients in the ICU
* Patients with hypoglycemic unawareness
* Outpatient insulin dose less than 0.6 units/kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-01-21 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Emanuele, MD, Principal Investigator — Loyola University
Locations (3):
- United States (3):
  - Northwestern University Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Hospital, Maywood, Illinois

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data available to other researchers

REFERENCES:
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. In 2007. Diabetes Care. 2008 Mar;31(3):596-615. doi: 10.2337/dc08-9017. PMID 18308683
- [Background] Baldwin D, Villanueva G, McNutt R, Bhatnagar S. Eliminating inpatient sliding-scale insulin: a reeducation project with medical house staff. Diabetes Care. 2005 May;28(5):1008-11. doi: 10.2337/diacare.28.5.1008. PMID 15855558
- [Background] DeSantis AJ, Schmeltz LR, Schmidt K, O'Shea-Mahler E, Rhee C, Wells A, Brandt S, Peterson S, Molitch ME. Inpatient management of hyperglycemia: the Northwestern experience. Endocr Pract. 2006 Sep-Oct;12(5):491-505. doi: 10.4158/EP.12.5.491. PMID 17002924
- [Background] Schmeltz LR, DeSantis AJ, Thiyagarajan V, Schmidt K, O'Shea-Mahler E, Johnson D, Henske J, McCarthy PM, Gleason TG, McGee EC, Molitch ME. Reduction of surgical mortality and morbidity in diabetic patients undergoing cardiac surgery with a combined intravenous and subcutaneous insulin glucose management strategy. Diabetes Care. 2007 Apr;30(4):823-8. doi: 10.2337/dc06-2184. Epub 2007 Jan 17. PMID 17229943
- [Background] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708
- [Background] Umpierrez GE, Hor T, Smiley D, Temponi A, Umpierrez D, Ceron M, Munoz C, Newton C, Peng L, Baldwin D. Comparison of inpatient insulin regimens with detemir plus aspart versus neutral protamine hagedorn plus regular in medical patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 Feb;94(2):564-9. doi: 10.1210/jc.2008-1441. Epub 2008 Nov 18. PMID 19017758
- [Background] Umpierrez GE, Smiley D, Jacobs S, Peng L, Temponi A, Mulligan P, Umpierrez D, Newton C, Olson D, Rizzo M. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes undergoing general surgery (RABBIT 2 surgery). Diabetes Care. 2011 Feb;34(2):256-61. doi: 10.2337/dc10-1407. Epub 2011 Jan 12. PMID 21228246
- [Background] Bernard JB, Munoz C, Harper J, Muriello M, Rico E, Baldwin D. Treatment of inpatient hyperglycemia beginning in the emergency department: a randomized trial using insulins aspart and detemir compared with usual care. J Hosp Med. 2011 May;6(5):279-84. doi: 10.1002/jhm.866. PMID 21661100
- [Background] Murad MH, Coburn JA, Coto-Yglesias F, Dzyubak S, Hazem A, Lane MA, Prokop LJ, Montori VM. Glycemic control in non-critically ill hospitalized patients: a systematic review and meta-analysis. J Clin Endocrinol Metab. 2012 Jan;97(1):49-58. doi: 10.1210/jc.2011-2100. Epub 2011 Nov 16. PMID 22090269
- [Background] Clement S, Braithwaite SS, Magee MF, Ahmann A, Smith EP, Schafer RG, Hirsch IB; American Diabetes Association Diabetes in Hospitals Writing Committee. Management of diabetes and hyperglycemia in hospitals. Diabetes Care. 2004 Feb;27(2):553-91. doi: 10.2337/diacare.27.2.553. No abstract available. PMID 14747243
- [Background] Moghissi ES, Korytkowski MT, DiNardo M, Einhorn D, Hellman R, Hirsch IB, Inzucchi SE, Ismail-Beigi F, Kirkman MS, Umpierrez GE; American Association of Clinical Endocrinologists; American Diabetes Association. American Association of Clinical Endocrinologists and American Diabetes Association consensus statement on inpatient glycemic control. Diabetes Care. 2009 Jun;32(6):1119-31. doi: 10.2337/dc09-9029. Epub 2009 May 8. No abstract available. PMID 19429873
- [Background] Umpierrez GE, Hellman R, Korytkowski MT, Kosiborod M, Maynard GA, Montori VM, Seley JJ, Van den Berghe G; Endocrine Society. Management of hyperglycemia in hospitalized patients in non-critical care setting: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2012 Jan;97(1):16-38. doi: 10.1210/jc.2011-2098. PMID 22223765
- [Background] Fischer KF, Lees JA, Newman JH. Hypoglycemia in hospitalized patients. Causes and outcomes. N Engl J Med. 1986 Nov 13;315(20):1245-50. doi: 10.1056/NEJM198611133152002. PMID 3534567
- [Background] Kagansky N, Levy S, Rimon E, Cojocaru L, Fridman A, Ozer Z, Knobler H. Hypoglycemia as a predictor of mortality in hospitalized elderly patients. Arch Intern Med. 2003 Aug 11-25;163(15):1825-9. doi: 10.1001/archinte.163.15.1825. PMID 12912719
- [Background] Varghese P, Gleason V, Sorokin R, Senholzi C, Jabbour S, Gottlieb JE. Hypoglycemia in hospitalized patients treated with antihyperglycemic agents. J Hosp Med. 2007 Jul;2(4):234-40. doi: 10.1002/jhm.212. PMID 17702035
- [Background] Turchin A, Matheny ME, Shubina M, Scanlon JV, Greenwood B, Pendergrass ML. Hypoglycemia and clinical outcomes in patients with diabetes hospitalized in the general ward. Diabetes Care. 2009 Jul;32(7):1153-7. doi: 10.2337/dc08-2127. PMID 19564471
- [Background] Bailon RM, Cook CB, Hovan MJ, Hull BP, Seifert KM, Miller-Cage V, Beer KA, Boyle ME, Littman SD, Magallanez JM, Fischenich JM, Harris JK, Scoggins SS, Uy J. Temporal and geographic patterns of hypoglycemia among hospitalized patients with diabetes mellitus. J Diabetes Sci Technol. 2009 Mar 1;3(2):261-8. doi: 10.1177/193229680900300206. PMID 20144357
- [Background] Rubin DJ, Rybin D, Doros G, McDonnell ME. Weight-based, insulin dose-related hypoglycemia in hospitalized patients with diabetes. Diabetes Care. 2011 Aug;34(8):1723-8. doi: 10.2337/dc10-2434. Epub 2011 Jun 23. PMID 21700919
- [Background] Horton ES, Johnson C, Lebovitz HE. Carbohydrate metabolism in uremia. Ann Intern Med. 1968 Jan;68(1):63-74. doi: 10.7326/0003-4819-68-1-63. No abstract available. PMID 5635331
- [Background] Moen MF, Zhan M, Hsu VD, Walker LD, Einhorn LM, Seliger SL, Fink JC. Frequency of hypoglycemia and its significance in chronic kidney disease. Clin J Am Soc Nephrol. 2009 Jun;4(6):1121-7. doi: 10.2215/CJN.00800209. Epub 2009 May 7. PMID 19423569
- [Background] Rave K, Heise T, Pfutzner A, Heinemann L, Sawicki PT. Impact of diabetic nephropathy on pharmacodynamic and Pharmacokinetic properties of insulin in type 1 diabetic patients. Diabetes Care. 2001 May;24(5):886-90. doi: 10.2337/diacare.24.5.886. PMID 11347749
- [Background] Mak RH. Impact of end-stage renal disease and dialysis on glycemic control. Semin Dial. 2000 Jan-Feb;13(1):4-8. doi: 10.1046/j.1525-139x.2000.00007.x. No abstract available. PMID 10740665
- [Background] Biesenbach G, Raml A, Schmekal B, Eichbauer-Sturm G. Decreased insulin requirement in relation to GFR in nephropathic Type 1 and insulin-treated Type 2 diabetic patients. Diabet Med. 2003 Aug;20(8):642-5. doi: 10.1046/j.1464-5491.2003.01025.x. PMID 12873291
- [Derived] Baldwin D, Zander J, Munoz C, Raghu P, DeLange-Hudec S, Lee H, Emanuele MA, Glossop V, Smallwood K, Molitch M. A randomized trial of two weight-based doses of insulin glargine and glulisine in hospitalized subjects with type 2 diabetes and renal insufficiency. Diabetes Care. 2012 Oct;35(10):1970-4. doi: 10.2337/dc12-0578. Epub 2012 Jun 14. PMID 22699288

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study took place at Loyola University Medical Center (Maywood, IL), Rush University Medical Center (Chicago, IL), and Northwestern University Medical Center (Chicago, IL) between January 2009 and May 2011
Groups:
- 0.5 Units/kg: Participants randomized to this arm receive a standard-dose of 0.5 units/kg daily insulin. Half of this dose is given as glargine and the other half as glulisine.
- 0.25 Units/kg: Participants randomized to this arm receive an experimental dose of 0.25 units/kg daily insulin. Half of this dose is given as glargine and the other half as glulisine.
Period: Overall Study
Arm/Group | 0.5 Units/kg | 0.25 Units/kg
Started | 57 | 57
Completed | 50 | 57
Not Completed | 7 | 0
Not completed — Lost to Follow-up | 7 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all patients who were randomized and completed all study activities
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 Units/kg | 0.25 Units/kg | Total
Number analyzed (Participants) | 50 | 57 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.6) | 63.7 (13.0) | 64.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 20 | 29 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 22 | 39
  White | 32 | 32 | 64
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73 squared meters] | 30.4 (8.3) | 29.6 (10) | 29.9 (9.0)
Years of Diabetes [Mean (Standard Deviation); unit: years] | 18.6 (8.8) | 16.6 (9.9) | 17.6 (10.0)
Glycated hemoglobin [Mean (Standard Deviation); unit: Percentage (%)] | 8.2 (2.1) | 7.9 (1.9) | 8.0 (2.0)
Insulin therapy before admission [Count of Participants; unit: Participants]
  Insulin before admission | 39 | 42 | 81
  No insulin before admission | 11 | 15 | 26
Total home daily insulin dose [Mean (Standard Deviation); unit: units of insulin] | 54.3 (40.7) | 51.6 (46.3) | 52.0 (43.0)

OUTCOME MEASURES:

1. Primary Outcome: Average Blood Glucose Over 6 Days
Description: Participants have their blood glucose measured daily for six days. The average blood glucose measure over all six days is compared between the two treatment cohorts.
Time Frame: 6 Days
Population: The analysis population for the primary outcome comprises all participants who were randomized and completed all study activities
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | 0.5 Units/kg | 0.25 Units/kg
Number analyzed (Participants) | 50 | 57
milligrams per deciliter | 174 (52.3) | 174.5 (46)
Statistical Analysis 1: Comparison: 0.5 Units/kg vs 0.25 Units/kg; The null hypothesis is that there is no difference between the two treatment cohorts on their average blood glucose level; Test type: Superiority; p = .958, t-test, 2 sided; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-19.341 to 18.341], Standard Error of Mean 9.502

2. Secondary Outcome: The Number of Participants Who Experience at Least One Blood Glucose Level Below 70 Milligrams Per Deciliter
Description: At the end of the study, the number of participants who experience at least one blood glucose level below 70 milligrams per deciliter (mg/dL) is compared between the two treatment cohorts
Time Frame: 6 Days
Population: This analysis comprises all participants who were randomized and completed all study activities
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 Units/kg | 0.25 Units/kg
Number analyzed (Participants) | 50 | 57
Participants
  At least one blood glucose level below 70 mg/dL | 15 | 9
  No blood glucose level below 70 mg/dL | 35 | 48
Statistical Analysis 1: Comparison: 0.5 Units/kg vs 0.25 Units/kg; The null hypothesis is that there is no difference in the odds of experiencing at least one blood glucose level below 70 mg/dL between the two treatment cohorts; Test type: Superiority; p = .0828, Regression, Logistic; Odds Ratio (OR) = 0.438, 95% CI 2-sided [0.172 to 1.114]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 years, 3 months
Arm/Group | 0.5 Units/kg | 0.25 Units/kg
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No